CLINICAL TRIAL: NCT00220688
Title: Does Acupressure Help Reduce Nausea and Vomiting in Palliative Care Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRC1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2007-03

CONDITIONS: Cancer
Keywords: nausea; vomiting; palliative; acupressure
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting

INTERVENTIONS:
Device: Acupressure Wristbands

SUMMARY:
Randomised controlled trial of acupressure wrist bands for hospice in-patients suffering from terminal cancer who are troubled by nausea and vomiting.

DETAILED DESCRIPTION:
Pilot The study will be piloted with 10 patients to ensure that the protocol is acceptable to patients and to inform a formal power calculation for a larger study. Patients will be randomized to each arm according to a randomization programme at www.randomization.com.

Arm 1 Instruction and placement of acupressure bands at the P6 acupuncture point bilaterally. This point is located 2 cun (a Chinese measurement equal to approximately 3cm) proximal to the midpoint of the transverse crease of the wrist between the tendons of palmaris longus and flexor carpi radialis.

Arm 2 Instruction and placement of sham acupressure bands P6 acupuncture point bilaterally. Sham acupressure bands have no stud to stimulate P6.

Patients may choose to have regular anti-emetics or a subcutaneous syringe driver after 24 hours if they are not happy with their level of nausea and vomiting.

4. STUDY POPULATION

4.1 Source and Number of Patients: Hospice in-patients. 10 patients for pilot.

4.2 Inclusion Criteria

Patients must meet the following criteria to be eligible to participate in the study:

1. Have a diagnosis of advanced cancer with an estimated prognosis of less than 1 year but more than 3 days.
2. Describe their nausea as at least moderate on a Likert scale OR at have had at least one vomit per day for the last three days.
3. Have an underlying cause for their nausea which is thought to be irreversible OR the patient has made an autonomous choice not to proceed with treatment for any potentially reversible cause (for example surgery for obstruction or drainage of ascites).
4. Can be male or female patients but must be over the age of 18.
5. Have signed a consent form prior to entering the study.
6. If patients are taking corticosteroids the dosage should be stable for 3 days before and during the trial.
7. Be thought to be well enough to complete the 3 day trial.

4.3 Exclusion criteria

1. Arm lymphoedema.
2. Weakness, fatigue or confusion sufficient that patient is unable to take part.
3. Previous history of acupuncture/acupressure for nausea or vomiting.
4. History of Parkinsonism or Parkinsonism on examination.
5. Patients will not be enrolled if they are sharing a room with another patient taking part in the study.

5. OUTCOME MEASURES

1. Visual Analogue Scale of nausea measured every 6 hours. If patients are asleep they will not be waken for assessments overnight.
2. Duration of perceived nausea over preceding time period.
3. Number of vomits per 24 hours.
4. Volume of vomit per 24 hours.
5. Adverse effects of acupressure.
6. Number of doses of PRN anti-emetics.
7. Measure of whether the patient felt the intervention helped at the end of the trial.

6. QUANTITATIVE ANALYSIS

This pilot will allow a formal power calculation to be performed to elucidate how many patients need to be randomized to the full study.

Statistical analysis will be performed by Sarah Vowler at the Centre for Applied Medical Statistics.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of advanced cancer with an estimated prognosis of less than 1 year but more than 3 days.
* Describe their nausea as at least moderate on a Likert scale OR at have had at least one vomit per day for the last three days.
* Have an underlying cause for their nausea which is thought to be irreversible OR the patient has made an autonomous choice not to proceed with treatment for any potentially reversible cause (for example surgery for obstruction or drainage of ascites).
* Can be male or female patients but must be over the age of 18.
* Have signed a consent form prior to entering the study.
* If patients are taking corticosteroids the dosage should be stable for 3 days before and during the trial.
* Be thought to be well enough to complete the 3 day trial.

Exclusion Criteria:

* Arm lymphoedema.
* Weakness, fatigue or confusion sufficient that patient is unable to take part.
* Previous history of acupuncture/acupressure for nausea or vomiting.
* History of Parkinsonism or Parkinsonism on examination.
* Patients will not be enrolled if they are sharing a room with another patient taking part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09; Study Completion 2006-10

PRIMARY OUTCOMES:
1.Visual Analogue Scale of nausea measured every 6 hours.

SECONDARY OUTCOMES:
Duration of perceived nausea over preceding time period.
Number of vomits per 24 hours.
Volume of vomit per 24 hours.
Adverse effects of acupressure.
Number of doses of PRN anti-emetics.
Measure of whether the patient felt the intervention helped at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perkins, MB BCh MRCP, Principal Investigator — Sue Ryder Care St. John's Hospice
Locations (1):
- Sue Ryder Care St. John's Hospice, Moggerhanger, Bedfordshire, United Kingdom

REFERENCES:
- [Result] Brown S, North D, Marvel MK, Fons R. Acupressure wrist bands to relieve nausea and vomiting in hospice patients: do they work? Am J Hosp Palliat Care. 1992 Jul-Aug;9(4):26-9. doi: 10.1177/104990919200900409. PMID 1457233